CLINICAL TRIAL: NCT04712253
Title: Multicenter Retrospective International Study to Evaluate Outcomes and Safety of Patients Undergoing ERCP Using a Single-use Cholangioscope (SpyGlass DS II) and Single-use Duodenoscope (Exalt) - The MESE Study
Brief Title: International Study to Evaluate Outcomes and Safety of Patients Undergoing ERCP Using a Single-use Cholangioscope and Single-use Duodenoscope
Acronym: MESE
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 101
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Biliary Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since its introduction more than 40 years ago, endoscopic retrograde cholangiopancreatography (ERCP) has fundamentally changed the treatment of biliopancreatic diseases. Since late 1970s there have been sporadic reports of nosocomial infections linked to endoscopic procedures, the majority caused by inadequate reprocessing of endoscopes. Infections due to multidrug-resistant organisms (MDROs) however have increasingly become a concern in health care, including in gastrointestinal (GI) endoscopy. Since 2010, reports of individual cases and serial outbreaks of MDRO infections associated with ERCP have been published worldwide. This is because, unlike a gastroscope or colonoscope, the duodenoscope is a complex instrument with unique mechanical features incorporated at the distal tip. This includes a recessed space containing an elevator, a wire cable that moves the elevator, working channel, and most recently, a seal that prevents contamination of the elevator wire channel. This complex design creates hard-to-reach areas that make optimal mechanical cleaning and disinfection difficult. With the aim of overcoming these issues, a single-use duodenoscope (EXALT Model D, Boston Scientific Corporation, Marlborough, Massachusetts, USA) has been developed in the United States of America (USA) and approved by the United States Food and Drug Administration (FDA) for clinical use in December 2019. Different studies evaluating this new device, including randomized clinical trials (RCTs), have already been published, which have confirmed that single-use duodenoscopes represent an alternative to reusable duodenoscopes for performing low-complexity ERCP procedures in experienced hands.

Digital Single Operator Cholangioscopy (D-SOC) using the single use Spyglass DS II (Boston Scientific Corporation, Marlborough, Massachusetts, USA) is a diagnostic and therapeutic modality which allows for direct endoscopic visualization of the biliopancreatic ductal system.

The principal diagnostic indication of D-SOC are bile duct or pancreatic strictures and unclear filling defects, adding direct endoscopic appearance data to biopsy sampling or brush cytology in order to improve the diagnostic yield.

The major therapeutic indication for D-SOC is lithotripsy for difficult biliary and pancreatic stones.

However, cholangioscopy increased the risk of post ERCP cholangitis. Bacteremia was suggested to be specifically related to cholangioscopy in 13.9% of 72 patients, based on serial blood samplings, and to be associated with biopsy sampling and strictures.

For this reason, the recent European Society of Gastrointestinal Endoscopy (ESGE) guideline suggests that patients should be considered to be at high risk for post-ERCP cholangitis when cholangioscopy is performed.

Presently, there are very few clinical reports about technical and clinical outcome of ERCPs performed with single use duodenoscope and there is complete lack of data about efficacy, safety and adverse events of the combination of the new single-use duodenoscope and the Spyglass DS II.

The aim of this multicentric retrospective study was to evaluate the technical success, clinical outcome and rate of adverse events of this procedure.

ELIGIBILITY:
Inclusion Criteria:

- patients that required an ERCP with cholangioscopy performed with the single-use EXALT duodenoscope in combination with the Spyglass DS II

Exclusion Criteria:

* Age < 18
* Lack of follow-up data (30 days at least)
* Less than 3 cases performed during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that required an ERCP with cholangioscopy performed with the single-use EXALT duodenoscope in combination with the Spyglass DS II between January 2020 and the time the IRB\Ethics Committee (EC) has approved the protocol for this retrospective series. The date of IRB\EC approval will vary from center to center. At each center, retrospective data collection will be completed immediately upon the local IRB\EC approval. The study plan is to complete the retrospective series by July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Technical success | 6 Months
  Technical success defined as the ability to successfully complete the entire procedure (completed without cross-over to a reusable duodenoscope) with the intended diagnostic or therapeutic maneuvers according to the clinical indication (i.e. stone fragmentation/removal, biopsies from the targeted tissue, etc)
Clinical Outcome | 6 Months
  Numbers of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No